CLINICAL TRIAL: NCT04753749
Title: Evaluation of a Modified Anti-Platelet Therapy Associated With Low-dose DES Firehawk in Acute Myocardial Infarction Patients Treated With Complete Revascularization Strategy
Acronym: TARGET-FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFHI01
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Infarction, Acute; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shortened DAPT followed by P2Y12 inhibitor monotherapy (Experimental)
  Interventions: Drug: Shortened DAPT followed by P2Y12 inhibitor monotherapy (cessation of aspirin)
- Dual Antiplatelet Therapy (Active Comparator)
  Interventions: Drug: Standard DAPT

INTERVENTIONS:
Drug: Shortened DAPT followed by P2Y12 inhibitor monotherapy (cessation of aspirin) — Subjects will receive DAPT during 1 month post procedure, followed by P2Y12 inhibitor monotherapy (cessation of aspirin) for the next 11 months
  Arms: Shortened DAPT followed by P2Y12 inhibitor monotherapy
Drug: Standard DAPT — Subjects will receive standard treatment: P2Y12 inhibitor and aspirin (DAPT) during 12 months after procedure
  Arms: Dual Antiplatelet Therapy

SUMMARY:
The study aims to evaluate a modified antiplatelet therapy associated with Firehawk low-dose rapamycin DES in acute myocardial infarction patients treated with complete revascularization strategy. The modified antiplatelet therapy consists of a reduced duration of Dual Antiplatelet Therapy post procedure (ie. 1 month duration) followed by P2Y12 inhibitor monotherapy for the next 11 months. It is hypothesized that in the setting of clinically stable, low to moderate complexity acute Myocardial Infarction patients, a modern approach combining a stent with high biocompatibility feature, complete revascularization strategy and modified antiplatelet therapy may be associated with similar outcomes, or even a significant benefit compared with guidelines-recommended 12-month DAPT. This benefit could be driven by a reduced risk in significant bleeding events, while keeping a comparable protection against ischemic risk. Enrolled subjects will be randomized in a 1:1 ratio to either cessation of aspirin at 1 months, either continuation of DAPT. Selection of the P2Y12 inhibitor agent is left to investigator judgment but has to be in line with the current ESC guidelines. Subjects treated with the Firehawk or Firehawk Liberty coronary stent will be included in this study.

ELIGIBILITY:
Inclusion Criteria (General):

* Troponin-positive Non-ST-Elevation MI, requiring early invasive treatment (PCI), or ST-Elevation MI requiring primary PCI, and PCI occurred within the last 7 days
* Subject is eligible for per-protocol antiplatelet treatments
* Written informed consent

Inclusion Criteria (Procedural/angiographic):

* Successful revascularization
* All treated lesions:

  * In native coronary arteries only
  * In vessels with visual reference diameter ≥2.25 mm and ≤ 4.00 mm
  * Implanted with the study device
  * Maximum 3 lesions treated (*)
  * Maximum total stent length ≤ 80 mm
* Complete revascularization performed when more than 1 significant lesion, during the index procedure or in staged procedure(s) occurring within 7 days from the index procedure.

Exclusion Criteria (General):

* Subjects with prior STEMI or prior PCI within 12 months before index admission
* Prior Coronary Artery Bypass Graft (CABG) Surgery
* Cardiogenic shock
* Secondary PCI
* Fibrinolysis
* Prior stent thrombosis
* Planned PCI, CABG, or surgery within 12 months
* Need for Oral Anti-Coagulation therapy
* Ischemic stroke or ICH within 12 months
* eGFR <30 mL/min/1.73 m2 or dialysis
* Active bleeding at time of inclusion or high risk for major bleeding
* History of bleeding diathesis or coagulopathy or subject refuse blood transfusions
* Stage B or C liver cirrhosis or active cancer within 12 months
* Baseline haemoglobin <13 g/dL (12g/dL for women) or anaemia requiring transfusion in the 4 weeks prior to index procedure
* Moderate or severe thrombocytopenia
* Expected non-adherence to protocol or estimated life expectancy ≤12 months
* Known hypersensitivity or contraindication to any medication used in the study or any of the study stent's components/compounds
* Participation in another interventional clinical trial
* Woman who is pregnant, nursing or with known intention to procreate

Exclusion Criteria (Procedural/Angiographic):

* In-stent restenosis or thrombosis
* Chronic total occlusion
* Severe calcification
* True bifurcation disease and side branch diameter ≥ 2mm, or bifurcation treated with 2 stents
* Left main coronary artery lesion
* Residual untreated dissection ≥ C
* Implantation of a non-study stent
* Subject is deemed to receive preferentially CABG within 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2248 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Net Adverse Clinical and Cerebral Events (NACCE) | 11 months post randomization
  (Number of participants with first occurrence of) NACCE, defined as a composite of all cause death, non-fatal myocardial infarction, definite/probable stent thrombosis, stroke, or bleeding events (BARC type 3 or 5)

SECONDARY OUTCOMES:
Bleeding events | 11 months post randomization
  (Number of participants with first occurrence of) bleeding events (BARC 2,3 or 5)
All-cause death, non-fatal myocardial infarction, definite/probable stent thrombosis, or stroke | At 1 month, 6 months and 12 months
  (Number of participants with first occurrence of) all-cause death, non-fatal myocardial infarction, definite/probable stent thrombosis, or stroke
Primary endpoint component 5 - BARC 3 and 5 bleeding events | At 1 month, 6 months and 12 months
  (Number of participants with first occurrence of) BARC 3 and 5 bleeding events
All-cause death or non-fatal myocardial infarction | At 1 month, 6 months and 12 months
  (Number of patients with first occurrence of) all-cause death or non-fatal myocardial infarction
Major Adverse Cardiac and Cerebral Events (MACCE) - Patient | At 1 month, 6 months and 12 months
  Patient-oriented composite of major adverse cardiac and cerebral events (MACCE) including all-cause death, myocardial infarction, definite/probable stent thrombosis, any stroke, any Ischemia driven repeat revascularization, or BARC bleeding events (type 2, 3, or 5)
Target Lesion Failure - Device | At 1 month, 6 months and 12 months
  Device oriented composite endpoint of Target Lesion Failure (cardiac death, target vessel related myocardial infarction, target lesion Ischemia Driven-revascularization)
Major Adverse Cardiac and Cerebral events (MACE) - Events | At 1 Month, 6 months and 12 months
  Number of Major Adverse Cardiac and Cerebral events (MACE)
Primary endpoint component 3 - Stent thrombosis | At 1 months, 6 months and 12 months
  Definite or probable stent thrombosis
Main secondary endpoint component 2 - BARC 3 events | At 1 month, 6 months and 12 months
  (Number of patients with occurrence of) BARC 3 events
Main secondary endpoint component 3 - BARC 5 events | At 1 month, 6 months and 12 months
  (Number of patients with occurrence of) BARC 5 events
Main secondary endpoint component 1 - BARC 2 events | At 1 month, 6 months and 12 months
  (Number of patients with occurrence of) BARC 2 events
Cardiovascular death | At 1 months, 6 months and 12 months
  Number of patients with cardiovascular death
Cardiac death | At 1 month, 6 months and 12 months
  Number of patients with cardiac death
Non cardiac death | At 1 month, 6 months and 12 months
  Number of patients with non cardiac death
Primary endpoint component 2 - Myocardial infarction | At 1 month, 6 months and 12 months
  Number of patients with myocardial infarction
Cardiac death or non-fatal myocardial infarction | At 1 month, 6 months and 12 months
  (Number of patients with first occurrence of) cardiac death or non-fatal myocardial infarction
Cardiac death, myocardial infarction, or definite/probable stent thrombosis | At 1 month, 6 months and 12 months
  (Number of patients with first occurrence of) cardiac death, myocardial infarction, or definite/probable stent thrombosis
Cardiovascular death, myocardial infarction, definite/probable stent thrombosis, or ischemic stroke | 1 month, 6 months and 12 months
  (Number of patients with first occurrence of) cardiovascular death, myocardial infarction, definite/probable stent thrombosis, or ischemic stroke
Primary endpoint component 4 - Ischemic stroke | At 1 month, 6 months and 12 months
  (Number of patients with occurrence of) ischemic stroke
Haemorrhagic stroke | At 1 month, 6 months and 12 months
  (Number of patients with occurrence of) haemorrhagic stroke
Ischemia-driven target lesion revascularization | At 1 month, 6 months and 12 months
  (Number of patients with) Ischemia-driven target lesion revascularization
Ischemia-driven target vessel revascularization | At 1 month, 6 months and 12 months
  (Number of patients with) Ischemia-driven target vessel revascularization
Cardiovascular death, myocardial infarction, or ischemic stroke | At 1 month, 6 months and 12 months
  (Number of patients with first occurrence of) cardiovascular death, myocardial infarction, or ischemic stroke
Primary endpoint component 1 - All cause death | At 1 month, 6 months and 12 months
  (Number of patients with) all cause death
Primary endpoint component 2 - Myocardial infarction | At 1 month, 6 months and 12 months
  (Number of patients with occurrence of) myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Tarantini, Pr, Principal Investigator — Padova University Hospital, Italy; Cayla Guillaume, Pr, Study Director — Nîmes University Hospital, France; Smits Peter, Pr, Study Director — Maastad University Hospital, Netherlands
Locations (40):
- Universitätsklinikum, Sankt Pölten, Austria
- France (20):
  - CHU Annecy, Annecy
  - Clinique Roseraie, Aubervilliers
  - CH Bastia, Bastia
  - CHU Caen, Caen
  - CH Chartres, Chartres
  - CH Cherbourg, Cherbourg
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CH Haguenau, Haguenau
  - CHU Lille, Lille
  - CH St Joseph/St Luc, Lyon
  - CHU La Timone, Marseille
  - Hôpital Jacques Cartier, Massy
  - CHU Montpellier, Montpellier
  - Clinique Millénaire, Montpellier
  - CHU Nîmes, Nîmes
  - CHU Reims, Reims
  - Clinique St Hilaire, Rouen
  - CHU Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
- Italy (6):
  - Humanitas - Gavazzeni, Bergamo
  - Clinica Montevergine, Mercogliano
  - Niguarda, Milan
  - AOU Federico II, Napoli
  - Policlinico Universitario, Padua
  - Giovanni Paolo II, Ragusa
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Tergooi MC, Blaricum
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Maastad University Hospital, Rotterdam
  - Haga Ziekenhuis, The Hague
- Hospital Santa Maria, Lisbon, Portugal
- Spain (7):
  - Hospital General Universitario, Alicante
  - Clinic Hospital Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Puerta del mar, Cadiz
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat
  - Hosp. Doctor Lucus Augusti, Lugo
  - Hospital Universitario La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarantini G, Smits PC, Lhermusier T, Honton B, Range G, Piot C, Lemesle G, Ruiz Nodar JM, Godin M, Madera Cambero M, Motreff P, Cuisset T, Bouchez D, Poezevara Y, Cayla G. A prospective study comparing short versus standard dual antiplatelet therapy in patients with acute myocardial infarction: design and rationale of the TARGET-FIRST trial. EuroIntervention. 2023 Jun 19;19(3):240-247. doi: 10.4244/EIJ-D-22-01006. PMID 36999409
- [Derived] Tarantini G, Honton B, Paradies V, Lemesle G, Range G, Godin M, Mangin L, Cuisset T, Ruiz-Nodar JM, Brugaletta S, Lhermusier T, Piot C, De Poli F, Macia JC, Motreff P, Madera-Cambero M, Beygui F, Riccini P, Ranc S, Oreglia JA, Vaquerizo B, Poezevara Y, Bouchez D, Smits PC, Cayla G; TARGET-FIRST Investigators. Early Discontinuation of Aspirin after PCI in Low-Risk Acute Myocardial Infarction. N Engl J Med. 2025 Nov 27;393(21):2083-2094. doi: 10.1056/NEJMoa2508808. Epub 2025 Aug 31. PMID 40888726